CLINICAL TRIAL: NCT06216145
Title: The Effect of the Formative Assessment Method Applied in the Fundamental of Nursing Course on Students' Knowledge, Skills and Self-Efficacy Levels
Brief Title: The Effect of the Formative Assessment Method Applied in the Fundamental of Nursing Course
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Rukiye Kokkiz, Research Assistant, Fenerbahce University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2023-20/2
Record Dates: First submitted 2023-12-25; First posted 2024-01-22 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Formative Evaluation; Nursing Skill

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Before the skills exam, the 'Self-Efficacy Survey in the Most Commonly Used Skill-Requiring Practices in Nursing' will be administered. Apart from the end-of-term skill exam, students will be given a different skill exam than the control group, in which they will not receive any grades. For applications requiring invasive interventions, a skill test will be administered in the laboratory.
  For applications that do not require invasive intervention, a skill test will be administered in the clinical environment. At the end of the semester, students will be asked to fill out the 'Self-Efficacy Survey in Practices Requiring the Most Commonly Used Skills in Nursing'. At the end of the semester, students will be evaluated with 2 skill applications and skill exam scores to be selected by written exam and lottery method.
  Interventions: Other: formative evaluation
- conrol group (Placebo Comparator): At the end of the fall semester midterm exam, the 'Self-Efficacy Survey in Practices Requiring the Most Commonly Used Skills in Nursing' will be administered. At the end of the semester, students will be asked to fill out the 'Self-Efficacy Survey in Practices Requiring the Most Commonly Used Skills in Nursing'. This scale will measure self-efficacy. At the end of the semester, students will be evaluated with 2 skill applications and skill exam scores to be selected by written exam and lottery method. With these exams, skills and theoretical knowledge will be measured.
  Interventions: Other: formative evaluation

INTERVENTIONS:
Other: formative evaluation — Before the skills exam, the 'Self-Efficacy Survey in the Most Commonly Used Skill-Requiring Practices in Nursing' will be administered. Apart from the end-of-term skill exam, students will be given a different skill exam than the control group, in which they will not receive any grades. For applications requiring invasive interventions, a skill test will be administered in the laboratory.
  For applications that do not require invasive intervention, a skill test will be administered in the clinical environment. At the end of the semester, students will be asked to fill out the 'Self-Efficacy Survey in Practices Requiring the Most Commonly Used Skills in Nursing'. At the end of the semester, students will be evaluated with 2 skill applications and skill exam scores to be selected by written exam and lottery method

SUMMARY:
In nursing education, the course where students encounter these gains for the first time and which forms the basis for other professional courses is generally the Nursing Fundamentals Course. In order to develop psychomotor skills within the scope of the Nursing Fundamentals Course, models are used to include practical studies in skill laboratories after the theoretical explanation of the course. Formative evaluation, one of the evaluation methods, is a process that provides clear feedback in teaching, regulates learning, and aims to improve the student's success in the educational outcome. The main purpose here is to review the learning and teaching process. Efforts are made to obtain feedback on situations that are disrupted in the learning-teaching process, incomplete learning, difficulties in learning, and situations in which improvement is needed. The feedback obtained in this evaluation is developmental for both the student and the instructor. Therefore, formative assessment is one of the important elements of reflective learning and teaching. With this research, students will be evaluated with a standard exam to determine whether they have achieved the expected proficiency levels in their knowledge and skills and whether the educational program has achieved its goals. This exam aims to measure students' self-efficacy by creating an example that can be used in other education and training institutions.

Students will be assigned to experimental and control groups by random route sampling method according to their internship locations.

A survey and a check-list for each nursing skill practice will be used in the research.

Self-Efficacy Survey in the Most Commonly Used Skill-Requiring Practices in Nursing; It will consist of 4 questions containing personal information and 6 questions listing nursing skills determined in line with the literature. Additionally, a check-list will be prepared for 6 nursing skills.

ELIGIBILITY:
Inclusion Criteria:

* Taking a nursing fundamentals course
* Volunteering to participate in the study
* Being over 18 years old

Exclusion Criteria:

* Dropping out of the fundamentals of nursing course
* Filling out forms incompletely

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-02-29 (Estimated); Primary Completion 2024-03-28 (Estimated); Study Completion 2024-05-29 (Estimated)

PRIMARY OUTCOMES:
self-sufficiency | 2 months
  As a result of the research, the self-efficacy result of the experimental group is lower than the control group.Self-efficacy is based on students' self-report in line with the survey created by the researcher.
skill grade | 2 months
  As a result of the research, the skill grade result of the experimental group is lower than the control group. Skill score will be measured by the checklist created by the instructor at the end of the course period.
information note | 2 months
  As a result of the research, the information note result of the experimental group is lower than the control group. The information grade will be measured by the survey prepared by the instructor at the end of the course period.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Istanbul, Üsküdar, Turkey (Türkiye)